CLINICAL TRIAL: NCT00272155
Title: Can Antibiotic Prescriptions in Respiratory Tract Infections be Improved? A Cluster Randomized Educational Intervention in General Practice
Brief Title: An Intervention to Reduce Inappropriate Prescriptions of Antibiotics for Respiratory Infections in General Practice
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Jorund Straand, Professor Md PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 850657
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2005-12

CONDITIONS: Respiratory Tract Infections; Anti-Bacterial Agents
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Early Intervention, Educational

INTERVENTIONS:
Behavioral: Educational intervention — Educational outreach visits to the CME-groups, work-shops, audit and feedback
Behavioral: Educational intervention program — The 433 recruited GPs had a total of 1336 717 office consultations of which 171 679 (12.8%) were RTIs encounters for 118 621 different patients. The GPs participated in peer continuing medical education (CME) groups in southern Norway. A multifaceted intervention was tailored, where key components were educational outreach visits to the CME-groups, work-shops, audit and feedback. Prescription Peer Academic Detailers conducted the educational outreach visits. During these visits, evidence-based recommendations of antibiotic prescriptions for RTIs were presented and software handed out for installation in participants PCs, enabling collection of prescription data. These data was linked to corresponding data from the Norwegian Prescription Database (NorPD). Main outcomes are baseline proportion of inappropriate antibiotic prescriptions for RTIs and change in prescription patterns compared to baseline one year after the initiation of the tailored pedagogic intervention.

SUMMARY:
This study will explore the possible effect of a tailored educational intervention towards general practitioners, in order to improve antibiotic prescriptions for respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner
* Specialist in general practice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118621 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in antibiotic prescription patterns for respiratory infections | 1 year
  From the 1.336.717 office consultations, main outcomes data (baseline proportion of inappropriate antibiotic prescriptions for RTIs and change in prescription patterns compared to baseline) was measured 1 year after the initiation of the tailored pedagogic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Svein Gjelstad, MD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Gjelstad S, Hoye S, Straand J, Brekke M, Dalen I, Lindbaek M. Improving antibiotic prescribing in acute respiratory tract infections: cluster randomised trial from Norwegian general practice (prescription peer academic detailing (Rx-PAD) study). BMJ. 2013 Jul 26;347:f4403. doi: 10.1136/bmj.f4403. PMID 23894178
- [Derived] Fossum GH, Lindbaek M, Gjelstad S, Dalen I, Kvaerner KJ. Are children carrying the burden of broad-spectrum antibiotics in general practice? Prescription pattern for paediatric outpatients with respiratory tract infections in Norway. BMJ Open. 2013 Jan 7;3(1):e002285. doi: 10.1136/bmjopen-2012-002285. PMID 23299114
- [Derived] Gjelstad S, Fetveit A, Straand J, Dalen I, Rognstad S, Lindbaek M. Can antibiotic prescriptions in respiratory tract infections be improved? A cluster-randomized educational intervention in general practice--the Prescription Peer Academic Detailing (Rx-PAD) Study [NCT00272155]. BMC Health Serv Res. 2006 Jun 15;6:75. doi: 10.1186/1472-6963-6-75. PMID 16776824